CLINICAL TRIAL: NCT02563470
Title: A Retrospective Registry of Bleeding, Cardio- and Cerebrovascular Complications in Patients Treated for Head and Neck Cancer
Brief Title: Bleeding, Cardio- and Cerebrovascular Complications in Head and Neck Surgery
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Tuomas Kiviniemi, Cardiologist, MD, PhD, University of Turku
Other Study IDs: HNS01
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this retrospective registry trial, the investigators sought to assess the incidence and predictors of cardiovascular and cerebrovascular complications as well as their derivatives (acute coronary syndrome, decompensated heart failure, an episode of atrial fibrillation requiring cardiologist consultation, stroke, pulmonary embolism and venous thromboembolism) in cohort of patients undergoing head and neck surgery.

DETAILED DESCRIPTION:
Inclusion criteria consisted of all the consecutive patients (n=456) diagnosed with head and neck cancer at Turku University Hospital between 1999 and 2008. Patients receiving palliative procedures were also included. Patients whose treatment had started in other institute or whose treatment was not finished in the investigators institute and patients with primary diagnosis of skin cancer were excluded from this study. All head and neck surgery operations (n=591) were assessed. Information was collected by the first author of this article from referral letters, patient files, anesthesiology reports, intensive care unit reports, laboratory database, radiology database, electrocardiograms and pathology reports. Death was certificated from national authority for collecting and compiling statistics on various fields of society and economy.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with head and neck cancer in Turku University hospital between 1999-2008

Exclusion Criteria:

* skin cancer, treatment started in other institute or not finished in our institute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: head and neck cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 5 years
myocardial infarction | 5 years
stroke | 5 years
bleeding | 30 days
decompensated heart failure | 5 years
new onset atrial fibrillation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Kiviniemi, MD, PhD, Study Director — Turku University Hospital